CLINICAL TRIAL: NCT06636604
Title: Development of a Decision Support Algorithm (DSA) for Detecting the Sciatic Nerve in Safe Injection Practices
Acronym: Nursiatic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IŞIK ATASOY
Record Dates: First submitted 2024-03-01; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Nurses; Injection Site; Sciatic Nerve; Pain; Satisfaction, Patient
Keywords: Nurse; Sciatic nerve; Decision support algorithm; Intramuscular injection; Pain; Satisfaction; Patients
MeSH Terms: conditions — Pain; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group: The effect of the decision support algorithm on pain and satisfaction during intramuscular injection will be examined.
  Interventions: Other: DSA(Decision Support Algorithm)
- Control Group (No Intervention): There is no intervention. Pain and satisfaction during intramuscular injection will be examined.

INTERVENTIONS:
Other: DSA(Decision Support Algorithm) — Intramuscular injection will be given to 30 volunteer patients using the decision support algorithm.
  Arms: Experimental Group

SUMMARY:
This project aims to develop an artificial intelligence-based decision support algorithm (DSA) for the detection of the sciatic nerve in safe intramuscular injection applications.

In the first phase of the project,developed an artificial intelligence-based decision support algorithm (DSA) for the detection of the sciatic nerve in safe intramuscular injection applications.

In the second phase of the project, with the integration of the Decision Support Algorithm (DSA) on a computer accompanied by a doctor and an engineer, the presence of the sciatic nerve was tested on 30 volunteers. The test resulted in achieving a 100% sciatic nerve image, confirming the reliability of the DSA.

Subsequently, information about the algorithm was provided to volunteers and nurses in the emergency department of Sakarya Training and Research Hospital who applied for intramuscular injection.

DETAILED DESCRIPTION:
This project aims to develop an artificial intelligence-based decision support algorithm (DSA) for the detection of the sciatic nerve in safe intramuscular injection applications.

Method This project was conducted between 01-05-2022 and 01-11-2023.

Data Collection Phase In the first phase of the project, approximately 1500 ultrasound images of the sciatic nerve were obtained from 50 volunteers in right and left positions. Subsequently, the sciatic nerve was labeled on these images. The dimensions of the collected data were normalized, noise reduction was applied, histogram equalization was performed, and class imbalance was addressed by balancing the data. The data were further augmented by applying techniques such as rotation, translation, reflection, and zooming. The YOLOv7 model was chosen for model selection. Parameter optimization was performed for YOLOv7, and preprocessing and data augmentation processes were completed for training the model. The hyperparameters of the YOLOv7 model were manually adjusted, followed by the use of automatic hyperparameter tuning tools, significantly enhancing the model's performance.

Integration and Testing Phase of the DSA In the second phase of the project, with the integration of the Decision Support Algorithm (DSA) on a computer accompanied by a doctor and an engineer, the presence of the sciatic nerve was tested on 30 volunteers subjects based on signals received through a USG probe.

Clinical Trial Phase Subsequently, information about the algorithm was provided to volunteers and nurses in the emergency department of Sakarya Training and Research Hospital who applied for intramuscular injection. Under the supervision of volunteer nurses, project coordinators, and researchers, injections were administered to 30 patients using the DSA and to 30 patients using the traditional method. After completing the injections, nurses filled out and signed the "System Usability Scale" (SUS). Additionally, the "Visual Pain Scale" and "Satisfaction Visual Scale for Injections" were used to assess patients' pain after the injection. Pain levels of volunteer patients were compared immediately after injection and 15 minutes later.

Keywords Nurse, sciatic nerve, decision support algorithm.

ELIGIBILITY:
Inclusion Criteria:

* The participant volunteered to take part in the research and is over 18 years of age.
* They have applied to the emergency department for an intramuscular injection and have not experienced any injection-related complications before.
* There is no risk of developing complications during the injection phase, such as bleeding, coagulation disorders, or drug allergy.
* Additionally, there is no scarring or abscess at the injection site.
* There should be no communication barriers, such as a psychological disorder or inability to speak Turkish.
* To participate in this study, it is necessary to be able to read and sign the informed consent form in Turkish.

Exclusion Criteria:

* Excluded were individuals who did not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain conditions of the patients after the injection will be determined. | Baseline
  The patient marks his or her pain on a 10 cm ruler, on one end of which the painlessness is written, and on the other end, the most severe possible pain is written.
Pain conditions of the patients after the injection will be determined. | 15 minutes
  The patient marks his or her pain on a 10 cm ruler, on one end of which the painlessness is

SECONDARY OUTCOMES:
The patients' satisfaction levels after the injection will be determined. | Baseline
  Visual Analog Scale (VAS) was used to evaluate the patients' satisfaction levels with the injection.
The patients' satisfaction levels after the injection will be determined. | 15 minutes
  Visual Analog Scale (VAS) was used to evaluate the patients' satisfaction levels with the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Işık ATASOY, MsC, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)